CLINICAL TRIAL: NCT06841224
Title: The Factors Affecting IPP in Peritoneal Dialysis Patients with Polycystic Kidney Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IPP in ADPKD
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Peritoneal Dialysis; Polycystic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Background: Polycystic kidney disease (PKD) is the most common hereditary kidney disease. Peritoneal dialysis (PD) in such patients is restricted because the significantly enlarged kidneys and liver may lead to the increase of intraperitoneal pressure (IPP). Increased IPP points to higher risk of abdominal wall complications and limited infusion volume that cause insufficient dialysis adequacy. Therefore, monitoring IPP is especially important in patients with polycystic kidney disease. However, the standard measurement of IPP is limited due to its cumbersome procedures, the application value of equation for estimating IPP among general peritoneal dialysis patients is not clear in the PKD population and the variables influence the IPP is yet to be explored..

Objective: The main purpose of our study was to validate the existing IPP equations in the PKD patients. Further, more relevant variables were included to optimize the IPP equation. Monitoring IPP can guide the formulation of peritoneal dialysis prescription for ADPKD patients, reduce the occurrence of abdominal wall complications, and the clinical utility and efficiency of PD was expanded.

Methods: A multi-center cross-sectional study. The IPPs were measured using the Durand method, with whole-body and abdominal anthropometry indices, the volume of abdominal cavity, the total kidney volume and liver volume were collected. New equation for estimate IPP in PKD patients were generated by stepwise linear regression modeling. The eIPP were calculated using two developed equations previously. Then The bias, accuracy and precision of eIPP derived from new equation were compared with actual IPP by Durand method respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years;
2. A confirmed diagnosis of polycystic kidney disease, with a history of peritoneal dialysis catheter placement and regular peritoneal dialysis;
3. Able to tolerate the infusion of more than 1500 mL of dialysis fluid.

Exclusion Criteria:

1. Acute complications such as peritonitis or cardiovascular and cerebrovascular events within the past month;
2. History of abdominal surgery or trauma within the past month;
3. History of kidney cyst rupture, infection, or bleeding within the past month;
4. History of abdominal or pelvic organ tumors;
5. History of abdominal pressure-related complications, such as hernias, leaks, or chest-abdominal fistulas;
6. Unable to attend follow-up visits during the study period;
7. Refusal to participate in the study. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 polycystic kidney disease patients undergoing peritoneal dialysis at 5-10 peritoneal dialysis centers nationwide from January 2024 to June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
intraperitoneal pressure | 20 minutes
  Actual IPP (aIPP) was measured as previously described by Durand et al.17. The peritoneal cavity was completely emptied before the test. The patient was placed briefly in a supine position on a horizontal plane and the height of the horizontal plane was standardized for all study subjects. A graduated column (cm) was bounded to the abdominal cavity through the PD catheter, with zero level placed on the midaxillary line. Two-liter dialysate solution was infused into the peritoneal cavity. We then read the height between the column of dialysate inside the PD catheter and the midaxillary line in centimetres of water (cmH2O) at non-deep expiration (IPP exp) and non-deep inspiration (IPP insp) respectively, calculating the mean of IPP exp and IPP insp. After outflowing 500 ml of the dialysate solution, we measured the aIPP again utilizing the same procedure. As a result, aIPP was measured two times for each participant. All the measurements were performed by two skillful nurses, which had

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university First hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data described in the manuscript, code book, and analytic code will not be made available because the Management of China's Human Genetic Resources.